CLINICAL TRIAL: NCT07263126
Title: Effect of Bicycle Ergometer Training in Thermoneutral and Lightly Cold Ambient Temperatures on Fat Tissue Amount and Metabolism in Overweight and Obese Women
Brief Title: Effect of Bicycle Ergometer Training on Fat Tissue Amount and Metabolism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Şule ŞİMŞEK, Principal İnvestigator, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23.07.2024/13
Record Dates: First submitted 2025-05-27; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Endurance Training
Keywords: Bicycle Ergometer; Overweight; Obese
MeSH Terms: conditions — Overweight; Obesity | interventions — Endurance Training

STUDY DESIGN:
Intervention Model Description: Endurance training in termoneutral ambient, Endurance training in lightly cold ambient, control group (the waiting list group)
Who Masked: Outcomes Assessor
Masking Description: The main outcome measures will be assessed by 3 different researchers . The researchers conducting the assessments will not know which group the participants are belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Case group 1 (Experimental): participants trained in termoneutral ambient temperature
  Interventions: Other: endurance training with bicycle ergometer in termoneutral ambient temperature
- Case group 2 (Active Comparator): participants trained in lightly cold ambient temperature
  Interventions: Other: endurance training with bicycle ergometer in lightly cold ambient temperature
- control group (No Intervention): participants do not trained

INTERVENTIONS:
Other: endurance training with bicycle ergometer in termoneutral ambient temperature — trained with bicycle ergometer three times a week for three months.
  Arms: Case group 1
Other: endurance training with bicycle ergometer in lightly cold ambient temperature — trained with bicycle ergometer three times a week for three months.
  Arms: Case group 2

SUMMARY:
The aim of this study is to investigate the effect of endurance training performed with a bicycle ergometer at different ambient temperatures on the amount of fat tissue and fat tissue metabolism in overweight and obese women.

DETAILED DESCRIPTION:
This study will examine the effects of 12 weeks of endurance training on a bicycle ergometer at thermoneutral and slightly cold ambient temperatures on body composition, subcutaneous and visceral fat tissue thickness, and levels of irisin, leptin, adiponectin, apelin, IL-6 and FGF-21 in the blood of overweight and obese women.

ELIGIBILITY:
Inclusion Criteria:

Being female,

* Being between 20-40 years old,
* Having a BMI between 25 and 34.9,
* Having a waist circumference greater than 80 cm,
* Not having participated in any exercise program in the last 3 months ,
* Not having experienced a change of more than 10% in body weight in the last 6 months.

Exclusion Criteria:

* On a weight loss diet,

  * Having cancer, unstable heart disease, cerebrovascular disease, metabolic disease, diabetes, hypertension, psychiatric disorders, or other conditions or neurological disorders,
  * Having a musculoskeletal disorder or any disease/injury that may affect participation in exercise training,
  * Participating in regular physical activity (at least 150 minutes of moderate-intensity physical activity or 75 minutes of vigorous-intensity physical activity or an equivalent combination of both during the week),
  * Being pregnant or breastfeeding,
  * Having undergone surgery for the treatment of obesity,
  * Receiving pharmacological treatment for obesity. Participants who did not attend more than 20% of the endurance training program will be excluded from the study.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-05-27 (Estimated); Study Completion 2026-05-27 (Estimated)

PRIMARY OUTCOMES:
rate of BMI | baseline/ through study completion, an average 3 months
  assesed with height and body weight
analysis of biyoelectric impedans Bioelectrical impedance analysis | baseline/ through study completion, an average 3 months
  assesed with with a Tanita BC 418 brand device.
Ratio of waist-hip Waist hip ratio | baseline/ through study completion, an average 3 months
  Waist and hip circumference will be measured with a tape measure.
rate of subcutaneous and visceral adipose tissue thickness | baseline/ through study completion, an average 3 months
  assesed with Ultrasonography
concentration of serum irisin, leptin, adiponectin, apelin, İL-6 and FGF-21 | baseline/ through study completion, an average 3 months
  assesed with blood analysis

CONTACTS AND LOCATIONS:
Overall Officials: Ummuhan Baş Aslan, Prof. Dr., Study Director — Prof. Dr.
Locations (1):
- Şule Şimşek, Denizli, Sarayköy, Turkey (Türkiye)

REFERENCES:
- [Result] Otero-Diaz B, Rodriguez-Flores M, Sanchez-Munoz V, Monraz-Preciado F, Ordonez-Ortega S, Becerril-Elias V, Baay-Guzman G, Obando-Monge R, Garcia-Garcia E, Palacios-Gonzalez B, Villarreal-Molina MT, Sierra-Salazar M, Antuna-Puente B. Exercise Induces White Adipose Tissue Browning Across the Weight Spectrum in Humans. Front Physiol. 2018 Dec 11;9:1781. doi: 10.3389/fphys.2018.01781. eCollection 2018. PMID 30618796